CLINICAL TRIAL: NCT00461136
Title: An Open-label, One-period, One-treatment Study to Evaluate the Time Course of the Antiproteinuric and Blood Pressure Lowering Effects After Initiation of Renin Inhibition With Aliskiren in Type 2 Diabetes Suffering From Incipient and/or Established Nephropathy
Brief Title: Time Course of the Antiproteinuric and Blood Pressure Lowering Effects After Initiation of Renin Inhibition With Aliskiren in Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A2242
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Type 2
Keywords: Time course; antiproteinuric; blood pressure; lowering effect; initiation of renin inhibition; Aliskiren in Type 2 diabetes; incipient and/or established nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
This study will evaluate the time-course of the antiproteinuric effect of renin inhibition with Aliskiren in patients with Type 2 diabetes suffering from incipient and/or established nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients from 30-80 years of age with a diagnosis of Type 2 diabetes (WHO criteria).
* Incipient and established diabetic nephropathy (urinary albumin excretion ≥ 100 mg/day but ≤ 2000 mg/day).
* Glomerular filtration rate (GFR) ≥ 40 ml/min (estimated using Modification of Diet in Renal Disease (MDRD) formula) in the last 4 months.
* Female patients must be postmenopausal or must have had a bilateral oophorectomy or must have been surgically sterilized or hysterectomized at least 6 months prior to screening.
* To be eligible patients must fulfill the following criteria: Patients on ongoing hypertensive therapy must have a blood pressure ≥ 135/85 mm Hg but lower than 170/105 mm Hg at baseline (Day -1) AND patients must be on stable antihypertensive medications for at least 8 weeks prior to baseline (Day -1).; Newly diagnosed hypertensive patients must have a blood pressure ≥ 135/85 mm Hg but lower than 170/105 mm Hg at baseline (Day -1).
* Patients must be on stable hypoglycemic medications for at least 8 weeks prior to Visit 2 ( Day -1).
* Patients must be willing and medically able to discontinue all Angiotensin-converting enzyme inhibitor (ACEI), Angiotensin receptor blocker (ARB), aldosterone receptor antagonist and potassium sparing diuretic medications for the duration of the study.
* Oral body temperature within the range 35.0-37.5 °C
* Able to provide written informed consent prior to study participation. .
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

* Severe Hypertension Grade 3 WHO classification (Mean Sitting Diastolic Blood Pressure (MSDBP) 110 mmHg and/or Mean Sitting Systolic Blood Pressure MSSBP 180 mmHg)
* Acetylsalicyclic acid (ASA) treatment >1g/day or regular use of Non steroidal anti-inflammatory drug (NSAIDs)
* Kidney disease not caused by diabetes or hypertension
* Serum potassium < 3.5 or > 5.1 mEq/L
* GFR < 40 ml/min/1.73m2 as measured by the MDRD formula
* Serum albumin < 2.0mg/dL
* History of hypertensive encephalopathy or cerebrovascular accident at any time prior to Visit1.
* Current diagnosis of heart failure (New York Heart Association (NYHA) Class II-IV)
* History of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any percutaneous coronary intervention (PCI) during the 6 months prior to Visit 1
* Second or third degree heart block without a pacemaker
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia
* Clinically significant valvular heart disease
* Type 1 diabetes mellitus
* Uncontrolled Type II diabetes mellitus (Hemaglobin subtype A1C (HbA1C) >11 %)
* History of malignancy including leukemia and lymphoma (but not basal cell skin carcinoma) within the past five years
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs including, but not limited to, any of the following:

History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection

-Currently active or previously active inflammatory bowel disease during the 12 months prior to Visit 1 Currently active gastritis, duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to Visit 1.

Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase Evidence of hepatic disease, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt

* Current treatment with cholestyramine or cholestipol resins
* History of immunocompromise, including a positive HIV test result.
* History of a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Persons directly involved in the execution of this protocol.
* Any condition that in the opinion of the investigator or the Novartis medical monitor would jeopardize the evaluation of efficacy or safety
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol
* Known or suspected contraindications to the study medications, including history of allergy to Angiotensin converting enzyme (ACE) inhibitors and/or to thiazide diuretics or other sulfonamide derived drug
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
* Use of any prescription drug or over-the-counter (OTC) medication which is prohibited by the protocol.
* Patients who previously participated in any Aliskiren study.
* Pregnant or nursing woman.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the time-course of the antiproteinuric effect of renin inhibition with Aliskiren in patients with Type 2 diabetes suffering from incipient and/or established nephropathy.

SECONDARY OUTCOMES:
To measure blood pressure changes over time during the onset and offset of effect.
To investigate whether there is a change on biomarkers of inflammation and cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis, Gentofte Municipality, Denmark